CLINICAL TRIAL: NCT03495011
Title: MRI Characterization of Mammographically Detected Calcifications and Ductal Carcinoma in Situ
Brief Title: MRI Characterization of Mammographically Detected DCIS
Status: Active, not recruiting | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 9778; R01CA203883 (NIH); RG3017004 (Other: Fred Hutch/University of Washington Cancer Consortium); NCI-2021-12034 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2018-04-04; First posted 2018-04-11 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer, Stage 0
Keywords: Ductal Carcinoma in Situ; MRI; Oncotype Dx
MeSH Terms: conditions — Breast Carcinoma In Situ; Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Cohort A: Patient with recently identified calcifications on mammography requiring biopsy. Patients will undergo a quantitative, multiparametric breast MRI as part of their clinical care. MRI will not change need for biopsy, but could identify additional suspicious sites. Only patients diagnosed with pure DCIS at biopsy and eventual surgical excision will receive Oncotype DX DCIS score testing.
  Interventions: Diagnostic Test: Breast MRI; Other: Laboratory Biomarker Analysis
- Cohort B: Patient with recent diagnosis of biopsy-proven DCIS would complete a research quantitative, multiparametric breast MRI as part of their clinical care. Only patients diagnosed with pure DCIS at surgical resection will receive Oncotype DX DCIS score testing.
  Interventions: Diagnostic Test: Breast MRI; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Diagnostic Test: Breast MRI — Quantitative, multiparametric breast MRI
Other: Laboratory Biomarker Analysis — Only patients with pure DCIS on surgical excision will have advanced pathologic markers and Oncotype Dx DCIS Score testing.
  Other Names: Oncotype Dx

SUMMARY:
This is a single institution, prospective observational clinical trial for women with mammographically identified calcifications that may represent ductal carcinoma in situ (DCIS).

The purpose of this study is to determine whether quantitative, multiparametric breast MRI performed prior to surgical resection can biologically characterize this common pre-invasive malignancy, ductal carcinoma in situ (DCIS), which typically presents in asymptomatic women as suspicious calcifications on mammography.

DETAILED DESCRIPTION:
The investigators will assess whether MRI signatures can determine which calcifications identified prior to surgical resection actually harbor DCIS, and whether these imaging features correlate with pathologic markers of proliferation (Ki-67) and inflammation (cox-2) within DCIS lesions.

The investigators will also explore whether quantitative MRI features in the peri-tumoral region correlate with prognostic microenvironment markers of inflammation (TNFα) and angiogenesis (VEGF). Finally, investigators will assess whether a multivariate model using these markers can accurately predict risk of recurrence based on a multi-gene assay (Oncotype DX DCIS score).

ELIGIBILITY:
Inclusion Criteria:

* [Cohort A] Women aged 18 or older with suspicious calcifications identified on mammography without an associated mass
* [Cohort B] Women aged 18 or older with recent biopsy-proven DCIS with residual calcifications present on mammogram after biopsy

Exclusion Criteria for Both Cohorts:

* Patients with prior history of breast cancer in the ipsilateral breast
* Patients with a newly diagnosed breast cancer in the contralateral breast
* Contra-indication to contrast-enhanced breast MRI (e.g. renal insufficiency with GFR<60, contrast allergy, incompatible metal)
* Patients who currently are undergoing chemoprevention therapy (e.g. aromatase inhibitors or selective estrogen receptor modulators)
* Women who are pregnant

Ages: 18 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Women aged 18 or older with suspicious mammographic caclifications or biopsy-proven DCIS with residual calcifications present on mammogram after biopsy. Study participants will undergo an experimental 3 Tesla breast MRI prior to surgical resection, including both DWI and DCE techniques. Only participants who are diagnosed with pure DCIS on both core needle biopsy and surgical resection will remain on study. Tissue from all DCIS lesions will also be sent for outside multi-gene assay testing (Oncotype DX DCIS score, Genomic Health, Redwood City, CA).
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2032-04 (Estimated)

PRIMARY OUTCOMES:
Fractional perfusion (f) | 3.5 years
  Assess whether high f within DCIS lesions correlates with proliferation (high Ki-67)
Tissue diffusion (Dt) | 3.5 years
  Assess whether low Dt within DCIS lesions correlates with high proliferation (Ki-67)
Transfer constant (Ktrans) | 3.5 years
  Assess whether high Ktrans within DCIS lesions correlates with inflammation (cox-2)

SECONDARY OUTCOMES:
Signal enhancement ratio (SER) | 3.5 years
  Assess whether low SER can exclude the presence of DCIS-associated malignancy at the site of mammographic calcifications
Apparent diffusion coefficient (ADC) | 3.5 years
  Assess whether high ADC can exclude the presence of DCIS-associated malignancy at the site of mammographic calcifications
Oncotype DCIS Score | 3.5 years
  Develop a multivariate MRI model to identify low risk DCIS (Oncotype DX DCIS score<39)
Transfer constant (Ktrans) | 3.5 years
  Assess whether high Ktrans in the peri-tumoral tissue correlates with stromal inflammation (TNFalpha)
Fractional perfusion (f) | 3.5 years
  Assess whether high f in the peri-tumoral tissue correlates with angiogenesis (VEGF)

CONTACTS AND LOCATIONS:
Overall Officials: Habib Rahbar, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No